CLINICAL TRIAL: NCT03213470
Title: Prospective Observation for Serial Changes in Acute Intracranial Artery Dissection Using High Resolution Vessel Wall Magnetic Resonance Imaging
Brief Title: Prospective Observation for Serial Changes in Acute Intracranial Artery Dissection Using HR-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Seung Chai Jung, MD. PhD., Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICD_01
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Arteries; Dissection
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

ARMS (1):
- Intracranial artery dissection (Other): Patients with intracranial artery dissection who were diagnosed based on the clinical and radiological (including MRI) diagnoses at the symptom onset after Jan-01-2016
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging

SUMMARY:
Intracranial artery disease has been more detected with development of HR-MR. HR-MR can depict vascular wall directly and give us more information beyond the pre-existing imaging modalities such as digital subtraction angiography, magnetic resonance angiography, computed tomography angiography. Hence, HR-MR is considered to become promising imaging modality for intracranial artery disease and many studies have been published recently. However, there was not enough to differentiate various intracranial artery disease such as atherosclerosis, dissection, moyamoya disease, vasculitis, reversible vasoconstriction syndrome. In real clinical arena, intracranial artery disease is too difficult to diagnose and distinguish among the disease. Of the disease, usefulness of HR-MR has been consistently published in the detection and diagnosis of intracranial artery dissection recently. HR-MR seems to be the most important and reliable imaging method in intracranial artery dissection as of now. Therefore, intracranial artery dissection is necessary to study using HR-MR. Intracranial artery dissection is dynamic vascular pathology. The geometric change is the most common among intracranial artery disease. However, there was no report about the geometric change in HR-MR. The investigators acquired retrospective data about the natural course of intracranial artery dissection in HR-MR and are preparing for publishing an article. However, the data is not prospective and not intraindividual comparison. Therefore, reliability is not enough to convince the natural course. If the investigators got prospective and intraindividual data, definite natural course of intracranial artery dissection could be acquired and would be helpful to diagnose the dissection and differentiate from other vascular pathologies. The longitudinal information from this study could guide us as the important map on the confusing HR-MR findings. In addition, the previous retrospective study can be a stepping-stone to perform a prospective study, which can increase the success rate of the prospective study. The protocols for imaging follow-up are as followed: initial (optional), 1 month, 3 month, 6 month (optional), 12 month

DETAILED DESCRIPTION:
Inclusion criteria:

1. adults with equal to or greater than 18 year-old
2. confirmed as acute intracranial artery dissection based on the clinical and radiological diagnoses
3. informed consent

Exclusion criteria:

1. contraindicated for MRI scanning and contrast media usage
2. refuse the enrollment

Outcome measures

1. Serial follow-up with intraindividual comparisons and interstage comparisons

   * Radiological features: intimal flap, double lumen, aneurysmal dilatation, intramural hematoma, luminal stenosis, contrast enhancement degree, diameters, length, wall thickness, eccentricity index
   * Clinical features: mRS, NIHSS, drug
2. Demographics

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Acute intracranial artery dissection

Exclusion Criteria:

* angioplasty, or stenting,
* contraindication for MR imaging,
* Hypersensitivity to gadolinium based contrast media,
* Pregnant or lactating women,
* Renal condition : eGFR < 60, 6) Patients unable and/or unwilling to comply with treatment or study instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2019-04-07 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
Prospective observation for serial changes in acute intracranial artery dissection using HR-MRI | The time interval from initial event to outcome measurement is 1 year.
  Radiological findings of HR-MRI during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Seung Chai Jung, Professor, Principal Investigator — Associate professor, Department of Radiology
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Park KJ, Jung SC, Kim HS, Choi CG, Kim SJ, Lee DH, Suh DC, Kwon SU, Kang DW, Kim JS. Multi-Contrast High-Resolution Magnetic Resonance Findings of Spontaneous and Unruptured Intracranial Vertebral Artery Dissection: Qualitative and Quantitative Analysis According to Stages. Cerebrovasc Dis. 2016;42(1-2):23-31. doi: 10.1159/000444315. Epub 2016 Mar 8. PMID 26950228
- [Derived] Jeong SY, Jung SC, Roh YH, Kwon SU, Kang DW, Kim JS, Choi KM, Kim S, Jeong E. Serial changes and optimal imaging windows in vessel wall MRI for unruptured intracranial artery dissection. Sci Rep. 2025 Jul 1;15(1):21864. doi: 10.1038/s41598-025-05732-4. PMID 40596300